CLINICAL TRIAL: NCT07195942
Title: Development of the Italian Version of the ICU Mobility Scale (IMS). Cross-cultural Adaptation, Italian Translation, and Validation Study.
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: IMS
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Muscle Weakness; Critical Illness; Critical Illness Recovery; Acquired Weakness
Keywords: Early Mobilisation; Muscle Weakness; Critical Illness; Acquired Weakness; Functional Mobility; Validation study; Inter-rater reliability
MeSH Terms: conditions — Muscle Weakness; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Early mobilisation of the patient admitted to intensive care units (ICUs) is essential to prevent Intensive Care Unit Acquired Weakness (ICUAW). It is essential to be able to measure functional mobility in order to evaluate the effectiveness of early mobilisation, both in clinical and research settings.

The ICU Mobility Scale (IMS) is a validated scale that can be used to describe the functional level of the critically ill patient according to a categorical scale of 11 items. Each category describes the patient's capabilities from a mobility point of view.

The main objective of the study is the validation of the Italian version of the IMS (IMS-it) on a cohort of patients admitted to intensive care.

Secondary objective is to assess the concordance between the perception level that the healthcare worker has with regard to the patient's mobility, before the patient is mobilised, expressed with the IMSSecondary study objectives.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 18 years
* ability self-mobility prior to hospital admission (assessed by the Clinical Frailty Scale), if applicable, the reasons for inclusion of vulnerable patients.

Exclusion Criteria:

* Concurrent admission due to newly diagnosed or suspected neurological disorders (e.g., stroke, intracranial hemorrhages, head trauma, Guillain-Barré syndrome, status epilepticus)
* Primary neurological or myopathic processes associated with muscle weakness (e.g. Guillain-Barré syndrome)
* Inability to understand and speak Italian
* History of cognitive deficits before hospital admission
* Unstable fractures or traumas requiring immobility, mobility restrictions, or bed rest
* Terminally ill patients in palliative care
* Any other clinical reasons that may prevent patient mobilization according to caring physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the General Intensive Care Unit (GICU) at the Humanitas Clinical Institute in Rozzano (MI)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Scale validity | From June 2023 to June 2025
  The correlation between IMS and other scales of muscular strength will be assessed using spearman correlation
Inter-rater reliability | From June 2023 to June 2025
  During the daily treatment of the patients by a healthcare professional, 1 critical care physiotherapist, 1 non-critical care physiotherapist and 1 critical care nurse will assess the patients enrolled in the study by means of the IMS.

SECONDARY OUTCOMES:
Predictive validity | From June 2023 to June 2025
  Correlation between IMS-it and clinical outcomes will be assessed, and adjusted through a multivariable logistic regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Greco, Anaesthesia and Intensive Care, Study Director — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Pieve Emanuele, Milano, Italy